CLINICAL TRIAL: NCT06987071
Title: Efficacy Of Acupuncture in Pain and Anxiety During Transperineal Prostate Biopsy: A Prospective, Randomized, Sham-Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ali Ihsan Memmi, MD, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 357843951
Record Dates: First submitted 2025-05-07; First posted 2025-05-23 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Pain Management; Acupuncture Analgesia; Prostate Biopsy
Keywords: acupuncture; prostate cancer; transperineal prostat biopsy; acupuncture anesthesia
MeSH Terms: conditions — Prostatic Neoplasms; Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, parallel-group trial. Participants are randomly assigned in a 1:1 ratio to receive either acupuncture or sham acupuncture 30 minutes prior to transperineal prostate biopsy. Both groups receive standard local anesthesia. Randomization is performed using a computer-generated sequence, and outcome assessors are blinded to group assignments.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Active Comparator): Participants receive acupuncture at specific points (LI4, PC6, ST36, SP6) for 20 minutes with manual stimulation, 30 minutes before the biopsy, alongside standard local anesthesia.
  Interventions: Procedure: Acupuncture
- Sham Acupuncture (Sham Comparator): Participants receive superficial needle insertion at non-acupuncture points without stimulation, 30 minutes before the biopsy, alongside standard local anesthesia.
  Interventions: Procedure: sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Insertion of sterile, single-use needles at specific acupuncture points (LI4, PC6, ST36, SP6) for 20 minutes with manual stimulation, administered 30 minutes before the biopsy by a licensed acupuncturist.
  Arms: Acupuncture
Procedure: sham acupuncture — Superficial needle insertion at non-acupuncture points without stimulation, administered 30 minutes before the biopsy, mimicking the acupuncture procedure without therapeutic intent.
  Arms: Sham Acupuncture

SUMMARY:
This randomized controlled trial evaluates the efficacy of acupuncture in reducing pain and improving patient experience during transperineal prostate biopsy. Participants will be randomized to receive either acupuncture or sham acupuncture prior to the biopsy, in addition to standard local anesthesia. The primary outcome is pain, measured using the Visual Analog Scale (VAS), while secondary outcomes include anxiety, additional analgesic use, patient satisfaction, and adverse events.

DETAILED DESCRIPTION:
Transperineal prostate biopsy is a standard diagnostic procedure for prostate cancer, often associated with pain and anxiety. Although local anesthesia is commonly used, it may not fully alleviate discomfort, and systemic medications can introduce side effects. Acupuncture, a traditional Chinese medicine technique, has demonstrated potential in managing procedural pain and reducing anxiety across various clinical settings. However, its specific efficacy for transperineal prostate biopsy remains underexplored.

This study aims to determine whether acupuncture, administered before the biopsy, can reduce pain, decrease anxiety, and enhance patient satisfaction compared to a sham procedure. Employing a randomized, single-blind design, the trial seeks to minimize bias and generate robust evidence regarding acupuncture's benefits in this context.

Participants will be randomly assigned to either the acupuncture group or the sham acupuncture group, with both receiving standard local anesthesia to ensure ethical care. Pain will be assessed using the Visual Analog Scale (VAS) at multiple time points, and anxiety will be measured with the State-Trait Anxiety Inventory (STAI). Additional outcomes include the use of supplementary analgesics, patient satisfaction, and any adverse events associated with the interventions.

The study's findings could inform clinical practice by introducing a complementary, non-pharmacological option for pain management during transperineal prostate biopsy, potentially improving patient comfort and reducing reliance on systemic medications.

The study protocol has been approved by the Institutional Review Board (IRB) of our hospital, and all participants will provide written informed consent prior to enrollment. Data will be collected and monitored by an independent data manager to ensure accuracy and patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for transperineal prostate biopsy (e.g., elevated PSA, abnormal digital rectal exam).
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Known allergy or contraindication to acupuncture (e.g., bleeding disorder, needle phobia).
* Requirement for sedation or general anesthesia.
* Previous experience with acupuncture treatment.
* Severe psychiatric disorders or diagnosed anxiety disorder.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Pain Score | Baseline, perioperative, 30 minutes post-biopsy, 2 hours post-biopsy.
  Visual Analog Scale (VAS), a 0-10 scale where 0 represents no pain and 10 represents the worst pain imaginable.

SECONDARY OUTCOMES:
Anxiety Level | before and after 30 minutes of operation
  State-Trait Anxiety Inventory (STAI), a validated questionnaire.
Additional Analgesic Use | after biopsy in 8 hours
  Type and dose of any additional pain medication required.
Adverse events | peri operative
  Any complications related to acupuncture or the biopsy procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Başakşehir Çam ve sakura City Hospita, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hong A, Hemmingway S, Wetherell D, Dias B, Zargar H. Outpatient transperineal prostate biopsy under local anaesthesia is safe, well tolerated and feasible. ANZ J Surg. 2022 Jun;92(6):1480-1485. doi: 10.1111/ans.17593. Epub 2022 Mar 10. PMID 35274426
- [Result] Yang J, Xiong X, Wei Q, Yang L. Acupuncture: a promising adjuvant strategy for pain management among the patients with prostate cancer. BJU Int. 2024 Oct;134(4):664-665. doi: 10.1111/bju.16467. Epub 2024 Jul 17. No abstract available. PMID 39019800
- [Result] Lin FX, Chen Y, Xu ZP. Enhancing perioperative pain management: the integrative potential of acupuncture in urological surgery. BJU Int. 2024 Oct;134(4):667-668. doi: 10.1111/bju.16503. Epub 2024 Aug 6. No abstract available. PMID 39106982
- [Result] Wang J, Lei Y, Bao B, Yu X, Dai H, Chen F, Li H, Wang B. Acupuncture for pain caused by prostate cancer: Protocol for a systematic review. Medicine (Baltimore). 2019 Jan;98(2):e13954. doi: 10.1097/MD.0000000000013954. PMID 30633174